CLINICAL TRIAL: NCT06042088
Title: Comparison of the Effect of Glove Number on Comfort, Sensitivity, and Dexterity in the Use of Double Surgical Gloves
Brief Title: Effect of Double Surgical Glove on Comfort, Sensitivity and Dexterity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Neslihan Ilkaz, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/170
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Surgical Gloves
Keywords: Surgical gloves; Comfort; Dexterity; Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Double Gloves:Regular Size (Experimental): Procedure A: Double gloves, participants will wear both gloves in their surgical glove size.
  Interventions: Other: Regular Size Glove and Bigger One
- Double Gloves: Regular Size and Half-Size Bigger (Experimental): Procedure B: Double gloves, Participants will wear their own glove size and half-size bigger glove on top
  Interventions: Other: Regular Size Glove and Bigger One
- Double Gloves: Half-Size Bigger and Regular Size (Experimental): Procedure C: Double gloves, participants will wear a half-size big glove and their own glove size on top.
  Interventions: Other: Regular Size Glove and Bigger One
- One Glove (No Intervention): Procedure D: Participants will wear only one glove.

INTERVENTIONS:
Other: Regular Size Glove and Bigger One — Different sizes of surgical gloves will be worn by participants
  Arms: Double Gloves: Half-Size Bigger and Regular Size; Double Gloves: Regular Size and Half-Size Bigger; Double Gloves:Regular Size

SUMMARY:
This clinical trial aims to test the effect of double surgical gloves worn in different sizes on the surgical team's comfort, sensitivity, and dexterity.

DETAILED DESCRIPTION:
The purpose of using surgical gloves is to create a protective barrier against blood-borne pathogens. According to studies, gloves can puncture during surgical procedures. Many studies recommend wearing double gloves. However, the World Health Organization reported that in the guideline for surgical site infections published in 2018, there is not enough evidence for wearing double or single gloves to prevent surgical site infections. However, he recommends that the surgical team prefer to use double gloves to protect themselves against punctures.

Although wearing double gloves is considered to be positive in terms of patient and employee safety, it is not preferred by the surgical team in some cases. The sense of touch and sensitivity of the human hand is at the center of surgical procedures. Finger pulp is extremely sensitive and contains many sensory receptors. Placing a barrier, such as a glove, between these sensory receptors and the touched surface may prevent tactile sensitivity in surgical applications. In addition to the advantages of double gloves in terms of patient and employee safety, there are disadvantages such as reduced dexterity and touch sensitivity. In the literature, it has been determined that there are few and old studies examining the effects of double glove use on performance and comfort. Therefore, this study, it was aimed to compare the effects of double surgical gloves worn in different procedures or usage habits (double gloves, large and small gloves) on the comfort, sensitivity, and dexterity of the surgical team.

The study will conduct as a prospective randomized controlled trial. After obtaining verbal and written consent from the participant, the study will conduct with various data collection forms. These forms are; the introductory information form, surgical glove evaluation form, and Visual Analogue Scale. Participants will randomize. After randomization, participants will be included in one of four groups. All procedures will be applied to participants in all groups. Group I (n=20), Group II (n=20), Group III (n=20), Group IV (n=20). Procedure A: Double gloves, participants will wear both gloves in their surgical glove size. Procedure B: Double gloves, participants will wear their own glove number and half a size bigger glove on top. Procedure C: Double gloves, participants will wear a half-size big glove and their own glove number on top. Procedure D: Participants will wear one glove (control procedure). Open surgeries with a duration of 90-120 minutes will be preferred for evaluation.

ELIGIBILITY:
Inclusion Criteria:

Taking part in the surgical team Six months or more of surgical experience

Exclusion Criteria:

Latex allergic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Change from comfort, sensitivity, and dexterity after 90-120 min. | After 90-120 minutes
  In this section, the degree of comfort, sensitivity, and dexterity. This status will be evaluated with Visual Analogue Scale. In Visual Analogue Scale we use between 0-10 point (0= most uncomfortable/ most insensitivity/ most indexterity, 10=most comfort/ most sensitivity/ most dexterity).

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Ilkaz, Principal Investigator — Ankara Medipol University
Locations (1):
- Neslihan Ilkaz, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Guo YP, Wong PM, Li Y, Or PP. Is double-gloving really protective? A comparison between the glove perforation rate among perioperative nurses with single and double gloves during surgery. Am J Surg. 2012 Aug;204(2):210-5. doi: 10.1016/j.amjsurg.2011.08.017. Epub 2012 Feb 17. PMID 22342011
- [Background] Bouvet E, Pellissier G, Abiteboul D, L'Heriteau F; Group for the Prevention of Occupational Infections in Healthcare Workers. Is double gloving an effective barrier to protect surgeons against blood exposure due to needlestick injury? Infect Control Hosp Epidemiol. 2009 Sep;30(9):928-9; author reply 929. doi: 10.1086/599309. No abstract available. PMID 19653826
- [Background] Schmauss D, Megerle K, Weinzierl A, Agua K, Cerny M, Schmauss V, Lohmeyer JA, Machens HG, Erne H. Microsurgeons do better--tactile training might prevent the age-dependent decline of the sensibility of the hand. J Peripher Nerv Syst. 2015 Dec;20(4):392-6. doi: 10.1111/jns.12144. PMID 26306813
- [Background] Mylon P, Carre MJ, Martin N, Lewis R. How do gloves affect cutaneous sensibility in medical practice? Two new applied tests. Proc Inst Mech Eng H. 2017 Jan;231(1):28-39. doi: 10.1177/0954411916679199. Epub 2016 Nov 23. PMID 27881806
- [Background] Global Guidelines for the Prevention of Surgical Site Infection. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK536404/ PMID 30689333
- [Background] Basak T, Sahin G, Demirtas A. Comparison of surgical gloves: perforation, satisfaction and manual dexterity. Int J Occup Saf Ergon. 2022 Jun;28(2):1160-1166. doi: 10.1080/10803548.2021.1875636. Epub 2021 Mar 2. PMID 33433290
- [Background] Han CD, Kim J, Moon SH, Lee BH, Kwon HM, Park KK. A randomized prospective study of glove perforation in orthopaedic surgery: is a thick glove more effective? J Arthroplasty. 2013 Dec;28(10):1878-81. doi: 10.1016/j.arth.2013.05.007. Epub 2013 Jun 6. PMID 23747130
- [Background] Moog P, Schulz M, Betzl J, Schmauss D, Lohmeyer JA, Machens HG, Megerle K, Erne HC. Do your surgical glove characteristics and wearing habits affect your tactile sensibility? Ann Med Surg (Lond). 2020 Aug 8;57:281-286. doi: 10.1016/j.amsu.2020.08.002. eCollection 2020 Sep. PMID 32904254
- [Background] Zhang Z, Gao X, Ruan X, Zheng B. Effectiveness of double-gloving method on prevention of surgical glove perforations and blood contamination: A systematic review and meta-analysis. J Adv Nurs. 2021 Sep;77(9):3630-3643. doi: 10.1111/jan.14824. Epub 2021 Mar 17. PMID 33733484
- [Derived] Parlak EA, Ilkaz N, Ayhan H, Iyigun E. Comparison of the effect of glove size on comfort, sensitivity and dexterity in the use of double surgical gloves: a randomized controlled trial. Int J Occup Saf Ergon. 2025 Jun 9:1-7. doi: 10.1080/10803548.2025.2503580. Online ahead of print. PMID 40485595